CLINICAL TRIAL: NCT06234397
Title: A Phase I, Open-Label, Multinational, Multicenter, Dose Escalation and Expansion Study of BH3120, as a Single Agent and in Combination With Pembrolizumab, in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation and Expansion Study of BH3120 Alone or With Pembrolizuamb in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-BAFP-101; KEYNOTE-F89 (Other: Merck Sharp & Dohme LLC); MK3475-F89 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BH3120 (Experimental): Arm A: BH3120 Monotherapy
  Interventions: Drug: BH3120
- BH3120 + pembrolizumab (Experimental): Arm B: BH3120 in combination with pembrolizumab
  Interventions: Drug: BH3120; Drug: pembrolizumab

INTERVENTIONS:
Drug: BH3120 — BH3120 will be administered as an IV infusion over 90 minutes on Day 1 of every 3-week treatment cycle
Drug: pembrolizumab — Fixed dose of pembrolizumab will be administered as an IV infusion over 30 minutes on Day 1 of every 3-week treatment cycle
  Other Names: KEYTRUDA®
  Arms: BH3120 + pembrolizumab

SUMMARY:
This is a First-in-Human, Phase 1, Dose-Escalation and Dose-Expansion study of BH3120, as a single agent and in combination with pembrolizumab, to assess safety, tolerability, MTD, RP2D, PK, and efficacy in patients with advanced or metastatic solid tumors. Dose-Escalation part is planned to establish the MTD or RD for Dose-Expansion part, while Dose-Expansion part is designed to assess potential efficacy of BH3120, as a single agent and in combination with pembrolizumab, when administered at the RD to subjects in indication-specific expansion cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a Histologically or cytologically confirmed non-CNS solid tumor that is metastatic or unresectable and for whom there is no available standard therapy.
* PD-L1 positive expression (Tumor Proportion Score ≥1% or Combined Positive Score ≥1).
* Have at least one lesion, not previously irradiated that can be accurately measured per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Age of 18 years or older (or country's legal age of majority if the legal age was >18 years)
* Adequate Hematologic and liver function.

Key Exclusion Criteria:

* Has received prior therapy with an anti-4-1BB(CD137) agent.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or has required active treatment.
* History of chronic liver disease or evidence of hepatic cirrhosis.
* History of severe toxicities associated with a prior immunotherapy.
* Has ongoing or suspected autoimmune disease.
* Known active and clinically significant bacterial, fungal or viral infection including known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, immunocompromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events and laboratory abnormalities graded per NCI-CTCAE v5.0. | Throughout the study until end of safety follow-up period (90 days after the last treatment)
  To evaluate safety and tolerability of BH3120 as a single agent and in combination with pembrolizumab administration
Incidence and nature of DLTs | At the end of Cycle 1 (each cycle is 21 days) in Dose-Escalation Part
  To evaluate safety and tolerability of BH3120 as a single agent and in combination with pembrolizumab administration

SECONDARY OUTCOMES:
The maximum serum concentration (Cmax) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The time to reach Cmax (Tmax) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The area under the concentration-time curve from time 0 to the last observable concentration (AUClast) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The AUC during the dosing interval (AUCtau) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The AUC extrapolated to infinity (AUCinf) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The terminal half-life (T1/2) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The apparent clearance (CL/F) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
The apparent volume of distribution (Vd/F) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon BH3120 administration
Frequency of anti-drug antibodies (ADA) | Throughout the study until treatment discontinuation (up to 2-3 years)
  Immunogenicity of BH3120
Objective response rate (ORR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  ORR will be measured as the proportion of subjects with a confirmed response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Disease Control Rate (DCR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  DCR will be measured as the proportion of subject with confirmed CR, PR, or Stable Disease (SD) as per RECIST v1.1
Duration of response (DOR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  DOR will be measured as the time from initial onset of CR or PR to first radiographic progression as per RECIST v. 1.1 or death from any cause, whichever occurs first.
Progression-free survival (PFS) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  PFS will be measured from date of first treatment until date of radiographic progression as per RECIST v.1.1 or until death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Carl & Edyth Lindner Center for Research & Education at The Christ Hospital and The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
  - Mays Cancer Center at University of Texas Health San Antonio MD Anderson Cencer Center, San Antonio, Texas
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul